CLINICAL TRIAL: NCT05223582
Title: Fluzoparib and Abiraterone in the preSurgery Treatment of Prostate Cancer: FAST Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAST trial
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: High-risk Prostate Cancer; Neoadjuvant Therapy
Keywords: Prostate cancer; Neoadjuvant therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; fluzoparib; Prednisone; Androgen Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib and abiraterone treatment group (Experimental): Patients would be treated with 1000mg abiraterone qd. Patients would be treated with 150mg fluzoparib bid. Patients would be treated with 5mg prednisone bid. Patients would get medical castration.
  Interventions: Drug: Abiraterone acetate; Drug: Fluzoparib; Drug: Prednisone; Drug: Androgen deprivation therapy; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Abiraterone acetate — Patients would be treated with 1000mg abiraterone qd.
Drug: Fluzoparib — Patients would be treated with 150mg fluzoparib bid.
Drug: Prednisone — Patients would be treated with 5mg prednisone bid.
Drug: Androgen deprivation therapy — Patients would get medical castration.
Procedure: Radical Prostatectomy — Patients would get radical prostatectomy after the neoadjuvant treatment.

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of fluzoparib combined with abiraterone in neoadjuvant treatment of patients with high-risk locoregional prostate cancer. Dr. Yao Zhu from Fudan University Shanghai Cancer Center is the co-leading PI of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Patients must have histologically or cytologically confirmed prostate adenocarcinoma, clinically assessed as localized or with only pelvic lymph node metastasis according to radiological evaluation, and categorized as high- or very-high risk per the National Comprehensive Cancer Network (NCCN) guidelines.
3. Patients need to maintain effective luteinizing hormone-releasing hormone analogue (LHRHa) therapy throughout the study treatment.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
5. Males choosing radical prostatectomy as the primary treatment for prostate cancer.
6. Normal bone marrow function: Absolute neutrophil count ≥ 1.5×10^9/L; platelets ≥ 100×10^9/L; hemoglobin ≥ 90g/L; white blood cell count ≥ 3.6×10^9/L.
7. Normal liver function: Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 ULN (upper limit of normal), total bilirubin ≤ 1.5 times ULN, Child-Pugh Class A, serum albumin ≥ 3g/dL.
8. Normal coagulation function: International normalized ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5 ULN, prothrombin time (PT) < ULN + 4 seconds.
9. Normal cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; QTc < 450ms for males, < 470ms for females, blood potassium ≥ 3.5mmol/L.
10. Normal blood pressure: Systolic blood pressure < 160mmHg, diastolic blood pressure < 95mmHg, patients with normal blood pressure after appropriate clinical treatment can be included.
11. Normal kidney function: Serum creatinine ≤ 1.5 ULN, creatinine clearance ≥ 50 mL/min.
12. Patients deemed to have the ability to ejaculate and an active sexual life must agree to use effective contraception and not to donate sperm from the first administration of the study drug until 3 months after the last administration.
13. Patients are able to understand and willing to sign the informed consent form. Patients are able to comply with the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patients with a history of other malignant tumors, myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML), or who have had other malignant tumors within 5 years before the first dosa (excluding completely resolved in situ cancers and malignancies deemed by the investigator to progress slowly).
2. Patients who have undergone local treatment for prostate cancer (such as radical prostatectomy, radiotherapy, or brachytherapy).
3. Patients who have received radiotherapy or major surgery within 3 weeks before the first dose or participated in another drug clinical trial within 4 weeks before the first dose.
4. Patients planning to receive any other antitumor therapy during the study treatment.
5. Patients who have received treatment with PARP inhibitors (e.g., fluzoparib, olaparib, talazoparib, veliparib, niraparib, lucaparib, or others), chemotherapy (e.g., docetaxel, cisplatin, carboplatin, oxaliplatin, or others), mitoxantrone, cyclophosphamide, CYP17 inhibitors such as ketoconazole, conventional anti-androgen therapy (luteinizing hormone-releasing hormone [LHRH] agonists/antagonists, bicalutamide, nilutamide), novel hormonal therapy (e.g., abiraterone, enzalutamide, apalutamide), or immunotherapy (e.g., sipuleucel-T vaccine, ipilimumab). Patients who have received conventional anti-androgen therapy or abiraterone for no more than 1 month are allowed to enroll.
6. Patients who have previous treated with strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, ritonavir, cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The washout period before the first dose should be at least 2 weeks.
7. Patients who have previous treated with strong CYP3A inducers (e.g., phenobarbital, phenytoin, rifampin, rifabutin, rifapentine, carbamazepine, nevirapine) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The washout period before the first dose should be at least 5 weeks for phenobarbital or enzalutamide and 3 weeks for other drugs.
8. Habitual drinking grapefruit juice or excessive tea, coffee, and/or caffeine-containing beverages, which cannot be discontinued during the study.
9. Inability to discontinue the use of medications that may affect P-glycoprotein (P-gp) during the study, including but not limited to amiodarone, carvedilol, clarithromycin, delavirdine, erythromycin, lapatinib, lopinavir, nelfinavir, propranolol, quinidine, ranolazine, tipranavir, and verapamil.
10. Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related diseases, active or symptomatic viral hepatitis, or chronic liver disease (HBV viral load ≥ 10^4 copies/mL, HCV viral load ≥ 10^3 copies/mL).
11. Clinically significant heart disease, such as New York Heart Association (NYHA) Class III-IV heart failure, myocardial infarction within the past 6 months, severe or unstable angina, or recent ventricular arrhythmias.
12. Preexisting duodenal stents or any gastrointestinal disorder or defect that the investigator believes would interfere with drug absorption.
13. Habitual constipation or diarrhea, irritable bowel syndrome, or inflammatory bowel disease; intra-abdominal fistula, gastrointestinal perforation, or abdominal abscess within the past 6 months, requiring blood transfusion for gastrointestinal bleeding.
14. Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors affecting medication intake and absorption.
15. History of asthma induced by nonsteroidal anti-inflammatory drugs (NSAIDs) or classified as "mild persistent" or more severe asthma history (symptoms ≥ 2 days per week).
16. History of uncontrolled pituitary or adrenal dysfunction, existing gonadal dysfunction, or severe hypogonadism.
17. Contraindications to the use of prednisone (corticosteroids) such as active infections or other lesions.
18. Any chronic disease requiring corticosteroid therapy at doses exceeding "prednisone 5mg, twice daily."
19. Allergy or intolerance to the active ingredients of fluzoparib, abiraterone, or prednisone.
20. History of neurological and psychiatric disorders such as dementia, epilepsy, or seizure susceptibility.
21. According to the investigator's judgment, there are severe concurrent diseases (such as severe diabetes, thyroid disease, and psychiatric illness, etc.) or unstable medical, psychological, or other conditions (including laboratory abnormalities) that may pose a serious risk to the subject's safety, affect the subject's completion of the study, or affect the study protocol and follow-up schedule.
22. Unsuitable for participation in this clinical trial for any reason according to the investigator's judgment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) or minimal residual disease (MRD) rate | 1 month after prostatectomy as local treatment for primary lesion
  Pathological response, defined as achieving either pCR or MRD at radical prostatectomy (RP). pCR is defined as the absence of morphologically identifiable carcinoma in the RP specimen. MRD will be defined as residual tumor in the RP specimen measuring ≤ 5 mm.

SECONDARY OUTCOMES:
Biochemical progression-free survival | Up to 2 years
Metastasis-free survival | Up to 2 years
PSA responses | During the treatment
surgical margins | 1 month after prostatectomy as local treatment for primary lesion
pathological stage | 1 month after prostatectomy as local treatment for primary lesion
radiological responses | 1 week before prostatectomy as local treatment for primary lesion
safety | During the treatment

OTHER OUTCOMES:
Prespecified and exploratory biomarkers | after prostatectomy as local treatment for primary lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD could be shared for scientific purposes by contacting the PI via email.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: The IPD could be shared for scientific purposes by contacting the PI via email.